CLINICAL TRIAL: NCT00282919
Title: A Phase 2, Open Label, Non-Comparative Trial Of Azithromycin 2000 mg Plus Chloroquine 600 Mg Base Daily For Three Days For The Treatment Of Uncomplicated Plasmodium Falciparum Malaria
Brief Title: A Three Day Trial of Azithromycin Plus Chloroquine for the Treatment of Uncomplicated Plasmodium Falciparum Malaria
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A0661154
Record Dates: First submitted 2006-01-26; First posted 2006-01-27 (Estimated); Results first posted 2014-06-26 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-05

CONDITIONS: Falciparum Malaria
MeSH Terms: conditions — Malaria, Falciparum | interventions — Azithromycin; Chloroquine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Azithromycin plus chloroquine (Experimental): Single Arm, Open label study
  Interventions: Drug: Azithromycin plus chloroquine

INTERVENTIONS:
Drug: Azithromycin plus chloroquine — dose of 2000 mg Azithromycin plus 600 mg chloroquine base

SUMMARY:
The treatment of symptomatic, uncomplicated malaria caused by P. falciparum in adults.

ELIGIBILITY:
Inclusion Criteria:

* Males and females greater then or equal to the age of 18 with uncomplicated, symptomatic malaria as indicated by the presence of blood smears positive for P. falciparum asexual parasitemia between 1000-100,000 parasites/uL and documented fever greater then or equal to 38.5 C/101.3 F rectal or fever greater then or equal to 38 C/100.4 F oral or history of fever as reported by subject within the prior 24 hours.

Exclusion Criteria:

* Subjects with severe or complicated malaria. Pregnant or breast feeding women.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2006-03; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- Pfizer Investigational Site, Tumaco, Departamento de Nariño, Colombia
- Pfizer Investigational Site, Bambolim, Goa, India

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0661154&StudyName=A%20Three%20Day%20Trial%20of%20Azithromycin%20Plus%20Chloroquine%20for%20the%20Treatment%20of%20Uncomplicated%20Plasmodium%20Falciparum%20Malaria%20

RESULTS

PARTICIPANT FLOW:
Groups:
- Azithromycin and Chloroquine: Four azithromycin 500 milligram (mg) tablets (equivalent to 2000 mg) orally once daily along with 2 chloroquine 300 mg base tablets (equivalent to 600 mg) orally once daily for 3 days.
Period: Overall Study
Arm/Group | Azithromycin and Chloroquine
Started | 110
Completed | 103
Not Completed | 7
Not completed — Lack of Efficacy | 4
Not completed — Withdrawal by Subject | 1
Not completed — Asymptomatic Parasitemia | 2

BASELINE CHARACTERISTICS:
Population: All treated population included participants who received at least 1 dose of study medication.
Arm/Group | Azithromycin and Chloroquine
Number analyzed (Participants) | 110
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.8 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25
  Male | 85

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Parasite Clearance at Day 28
Description: Parasite clearance was defined as the clearance of asexual Plasmodium falciparum (P falciparum) parasitemia (defined as three consecutive 0 parasite counts) within 7 days of initiation of treatment, without subsequent recrudescence up to Day 28. Failure to achieve clearance of asexual P falciparum parasitemia was defined as parasitemia not cleared within 7 days of initiation of treatment, or subsequent recrudescence (confirmed by molecular testing) by Day 28 after achieving clearance. Percentage of participants with clearance is reported. Here "N" (Number of participants analyzed) signify participants who were evaluable (parasitological per protocol) at Day 28.
Time Frame: Day 28
Population: Parasitological per protocol (PP) population: Participants who had study drug for 3 days unless treatment failure, no concomitant anti-malarial unless designated treatment failure, had test of cure at Day 28, baseline smear with parasitemia between 1000-100000 parasites/microliter, rapid diagnostic test positive for P falciparum, history of fever.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Azithromycin and Chloroquine
Number analyzed (Participants) | 107
percentage of participants | 97.20 [94.09 to 100.00]

2. Secondary Outcome: Percentage of Participants With Early Treatment Failures (ETF)
Description: ETF was defined as a participant meeting any of these criteria: development of signs of severe malaria (impaired consciousness [for example, obtundation, unarousable coma, delirium, stupor], respiratory distress [respiratory rate greater than or equal to {>=} 30 breaths/minute], seizures, hypoglycemia [glucose less than or equal to {<=} 40 milligram/deciliter], gross hematuria, increase in parasitemia to greater than 100,000 parasites/microliter in 48 hours or later after the first treatment dose was administered) any day from Day 0 to 3 in the presence of P falciparum parasitemia; parasite count on Day 2 > Day 0 (baseline), irrespective of axillary or oral temperature; parasite count on Day 3 > 37.5 degrees Celsius (axillary temperature) and >38 degrees Celsius (oral temperature) and parasite count on Day 3 >=25 percent (%) of the first available parasite density on Day 0 (baseline).
Time Frame: Baseline up to Day 28
Population: Parasitologic PP population. Here, "N" (Number of participants analyzed) signifies those who were evaluable for this outcome measure.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Azithromycin and Chloroquine
Number analyzed (Participants) | 107
percentage of participants | 0 [-0.47 to 0.47]

3. Secondary Outcome: Percentage of Participants With Late Treatment Failures (LTF)
Description: LTF included late clinical failure (LCF) and late parasitologic failure (LPF). LCF is defined as a participant meeting any of these criteria: development of signs or symptoms of severe malaria after Day 3 in the presence of P falciparum parasitemia, without previously meeting any of the criteria of ETF or presence of P falciparum parasitemia and fever or history of fever on any day from Day 4 to Day 28, without previously meeting any of the criteria of ETF. LPF is defined as presence of P falciparum parasitemia on any day from Day 7 to Day 28 and the absence of fever or history of fever without previously meeting any of the criteria of ETF or LCF.
Time Frame: Baseline up to Day 28
Population: as for outcome 2
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Azithromycin and Chloroquine
Number analyzed (Participants) | 107
percentage of participants | 2.80 [-0.3 to NA] — The upper limit of 90% CI was not estimable because very few participants had response.

4. Secondary Outcome: Percentage of Participants With Resistance to Treatment
Description: Resistance is measured by clearance of asexual P falciparum parasitemia and categorized into 3 levels; resistance I (RI): clearance of asexual P. falciparum parasitemia before Day 7 followed by recurrence on or after Day 7, resistance II (RII): marked reduction (<=25% of baseline) of asexual P. falciparum parasitemia but no clearance prior to and up to Day 7, and resistance III (RIII): no marked reduction (>25% of baseline) of asexual P. falciparum parasitemia. Recurrence was defined as the reappearance of asexual P. falciparum parasitemia following a quiescent or latent period after the cessation of the primary attack. Percentage of participants with resistance as measured by RI, RII and RIII is reported.
Time Frame: Days 7, 14, 21, 28, 35, 42
Population: Parasitologic PP population. Here, "N" (Number of participants analyzed) signifies those who were evaluable for this outcome measure and "n" signifies number of participants who were evaluated at given time point.
Measure: Number; unit: percentage of participants
Arm/Group | Azithromycin and Chloroquine
Number analyzed (Participants) | 109
percentage of participants
  Day 7 (n=109) | 22.02
  Day 14 (n=109) | 22.02
  Day 21 (n=107) | 22.43
  Day 28 (n=107) | 24.3
  Day 35 (n=107) | 25.23
  Day 42 (n=107) | 25.23

5. Secondary Outcome: Percentage of Participants With Clinical Cure
Description: Clinical Cure is defined as resolution of the participant's fever and other symptoms attributed to P falciparum malaria (for example, abdominal pain, malaise, and headache).
Time Frame: Day 3, 7, 28, and 42
Population: as for outcome 2
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Azithromycin and Chloroquine
Number analyzed (Participants) | 109
percentage of participants
  Day 3 | 100.00 [99.54 to 100.0]
  Day 7 | 100.00 [99.54 to 100.0]
  Day 28 | 96.33 [92.90 to 99.77]
  Day 42 | 96.33 [92.90 to 99.77]

6. Secondary Outcome: Percentage of Participants With Parasite Clearance at Day 7, 14, 21, 35, 42
Description: as for outcome 1
Time Frame: Day 7, 14, 21, 35, 42
Population: Parasitologic PP population. Here, "N" (Number of participants analyzed) signifies those participants who were evaluable for this outcome measure and "n" signifies number of participants who were evaluated at given time point.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Azithromycin and Chloroquine
Number analyzed (Participants) | 109
percentage of participants
  Day 7 (n=109) | 100.00 [99.54 to 100.00]
  Day 14 (n=109) | 100.00 [99.54 to 100.00]
  Day 21 (n=107) | 99.07 [97.06 to 100.00]
  Day 35 (n=107) | 96.26 [92.76 to 99.76]
  Day 42 (n=107) | 96.26 [92.76 to 99.76]

7. Secondary Outcome: Percentage of Participants With Gametocyte Clearance
Description: Gametocyte clearance was defined as clearance of P falciparum gametocytemia (defined as attainment of 3 consecutive 0 gametocyte counts) without subsequent recurrence through the day of consideration. Recurrence was defined as the reappearance of asexual P. falciparum gametocytemia after achieving clearance. Percentage of participants with gametocyte clearance were reported.
Time Frame: Day 7, 14, 21, 28, 35, 42
Population: as for outcome 4
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Azithromycin and Chloroquine
Number analyzed (Participants) | 109
percentage of participants
  Day 7 (n=109) | 84.40 [78.20 to 90.61]
  Day 14 (n=109) | 81.65 [75.07 to 88.24]
  Day 21 (n=106) | 77.35 [70.17 to 84.55]
  Day 28 (n=105) | 76.19 [68.84 to 83.54]
  Day 35 (n=103) | 76.69 [69.33 to 84.07]
  Day 42 (n=104) | 76.92 [69.61 to 84.23]

8. Secondary Outcome: Fever Clearance Time
Description: Fever clearance time (FCT) was defined as the time from baseline to the first of 2 consecutive time points with temperature less than (<) 37.5 degree Celsius (C) (axillary temperature) or <38 degree C (oral temperature).
Time Frame: Baseline up to Day 42
Population: Data not possible to report, as clearance time was obtained as life table plots only, as per planned analysis.
Arm/Group | Azithromycin and Chloroquine
Number analyzed (Participants) | 0

9. Secondary Outcome: Parasite Clearance Time
Description: Asexual P falciparum parasite clearance time was defined as the time from baseline to the first of the 3 consecutive 0 parasite counts.
Time Frame: Baseline up to Day 42
Population: Data not possible to report, as clearance time was obtained as life table plots only, as per planned analysis.
Arm/Group | Azithromycin and Chloroquine
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Azithromycin and Chloroquine
Serious Adverse Events (participants affected / at risk) | 0/110
Other Adverse Events (participants affected / at risk) | 54/110
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Azithromycin and Chloroquine (N=110)
Anaemia (Blood and lymphatic system disorders) | 1
Tachycardia (Cardiac disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 13
Gastritis (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 36
Vomiting (Gastrointestinal disorders) | 22
Pain (General disorders) | 1
Vaginitis bacterial (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Vulvovaginal candidiasis (Infections and infestations) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 6
Back pain (Musculoskeletal and connective tissue disorders) | 2
Depressed mood (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.